CLINICAL TRIAL: NCT02702193
Title: Set-Enhanced Aftercare for Mothers in Substance Abuse Recovery and Their Children
Brief Title: SET-Recovery/Healthy Home
Acronym: SET-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Victoria Mitrani, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20111132; U54MD002266 (NIH)
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Results first posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-11

CONDITIONS: Substance-Related Disorders; Mental Health
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SET-R/Healthy Home (Experimental): SET is a manualized, strength-based,directive and process-oriented family-ecosystemic intervention based on Brief Strategic Family Therapy. Healthy Home is an adaptation of SET to be delivered by nurses as an enhanced, family-strengthening, home-health intervention. Healthy Home is delivered in addition to the usual substance abuse or mental health outpatient services received by the mothers.
  Interventions: Behavioral: SET-R/Healthy Home
- TAU (No Intervention): Treatment as usual - the usual outpatient substance abuse or mental health services received by the mothers with no additional services provided by the study team.

INTERVENTIONS:
Behavioral: SET-R/Healthy Home — SET is a manualized, strength-based,directive and process-oriented family-ecosystemic intervention based on Brief Strategic Family Therapy. Healthy Home is an adaptation of SET to be delivered by nurses as an enhanced, family-strengthening, home-health intervention. Healthy Home is delivered in addition to the usual substance abuse or mental health outpatient services received by the mothers. The time-frame for the intervention is approximately 4 months, with home visits approximately every 2 weeks.
  Arms: SET-R/Healthy Home

SUMMARY:
The study conducts a community-based randomized trial comparing an adaptation of Structural Ecosystems Therapy (SET), "Healthy Home", as an enhancement of substance abuse or mental health outpatient treatment, to outpatient treatment as usual (TAU) among approximately 172 Black, Hispanic and White nonHispanic mothers enrolled in outpatient substance abuse or mental health services. The study is conducted with a community partner, Banyan Health Systems, that delivers substance abuse/mental health treatment and primary care. Data is collected at baseline and 4, 8, and 12 months postrandomization. The Specific Aims of the proposed study are to: 1) test the effectiveness of Healthy Home for improving physical and mental health and reducing relapse of mothers in substance abuse/mental health recovery; 2) test the effectiveness of Healthy Home for improving health and mental health outcomes of children of mothers in recovery; 3) test mechanisms of action of Healthy Home (self care, environmental risk, family functioning and stigma); 4) assess implementation and sustainability factors and the relationship between fidelity and outcomes; and 5) examine the interactions of ethnicity and ethnicity related factors on outcomes. Healthy Home is a manualized, strength-based, directive and process oriented family ecosystemic home health intervention developed to address the needs of mothers and their children affected by substance abuse and other mental health disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in outpatient substance abuse or mental health treatment (or treatment for substance abuse as a co-occurring disorder) or case management for mental health or substance abuse problems,
2. have at least one child age 0-17 with whom she has at least monthly contact
3. be age 18 or above,
4. capable of giving informed consent and comprehending either English or Spanish,
5. willing and able to participate fully in the protocol

Exclusion Criteria:

Persons who do not meet the inclusion criteria listed above will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The researcher will abide by NIH standards for sharing research resources developed through the study. Data will be made available no later than the date when the main findings are published. Upon request, electronic copies will be provided to researchers, along with data documentation. Data will not contain any personal identifiers. Researchers using these data will be asked to sign a data sharing agreement approved by the University of Miami. The primary purpose of this agreement will be to ensure that researchers using the dataset are aware of the potential risks to vulnerable groups, and take adequate protective steps.

REFERENCES:
- [Background] Mitrani VB, McCabe BE, Robinson C, Weiss-Laxer NS, Feaster DJ. Structural Ecosystems Therapy for recovering HIV-positive women: child, mother, and parenting outcomes. J Fam Psychol. 2010 Dec;24(6):746-55. doi: 10.1037/a0021638. PMID 21171773
- [Background] Feaster DJ, Burns MJ, Brincks AM, Prado G, Mitrani VB, Mauer MH, Szapocznik J. Structural Ecosystems Therapy for HIV+ African-American women and drug abuse relapse. Fam Process. 2010 Jun;49(2):204-19. doi: 10.1111/j.1545-5300.2010.01318.x. PMID 20594207
- [Background] Feaster DJ, Mitrani VB, Burns MJ, McCabe BE, Brincks AM, Rodriguez AE, Asthana D, Robbins MS. A randomized controlled trial of Structural Ecosystems Therapy for HIV medication adherence and substance abuse relapse prevention. Drug Alcohol Depend. 2010 Oct 1;111(3):227-34. doi: 10.1016/j.drugalcdep.2010.04.017. Epub 2010 Jun 9. PMID 20538417
- [Derived] Matsuda Y, McCabe BE, Behar-Zusman V. Mothering in the Context of Mental Disorder: Effect of Caregiving Load on Maternal Health in a Predominantly Hispanic Sample. J Am Psychiatr Nurses Assoc. 2021 Sep-Oct;27(5):373-382. doi: 10.1177/1078390320907693. Epub 2020 Feb 26. PMID 32102585

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening: 243 were screened of which there were 70 excluded (9 did not meet inclusion criteria; 32 declined participation; 29 were lost contacts)
Groups:
- Treatment As Usual (TAU): Treatment as usual - the usual outpatient substance abuse or mental health services received by the mothers with no additional services provided by the study team.
Period: Baseline Assessment/Randomization
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Started | 86 | 87
Completed | 85 | 87
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: 4 Month Follow up
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Started | 86 | 87
Completed | 68 | 69
Not Completed | 18 | 18
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 17 | 18
Period: 8 Month Follow up
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Started | 86 | 87
Completed | 71 | 69
Not Completed | 15 | 18
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 14 | 18
Period: 12 Month Follow up
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Started | 86 | 87
Completed | 69 | 69
Not Completed | 17 | 18
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SET-R/Healthy Home | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 85 | 87 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 87 | 172
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 87 | 172
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 65 | 72 | 137
  Race/Ethnicity: Black | 13 | 9 | 22
  Race/Ethnicity: White Non Hispanic | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Trajectory of Depression of Participants
Description: Self-reported experience with depressive symptoms as measured by the PROMIS depression scale over the past 7 days. Each item is scored 1-5 (1 = Never; 5 = Always), yielding a total between 8 and 40.
Time Frame: baseline, 4, 8 and 12 months
Population: Intent to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Number analyzed (Participants) | 85 | 87
Participants
  Participants Above Clinical Cutoff: Baseline | 40 | 28
  Participants Above Clinical Cutoff: 4 month | 18 | 27
  Participants Above Clinical Cutoff: 8 month | 25 | 23
  Participants Above Clinical Cutoff: 12 month | 21 | 23
Statistical Analysis 1: Comparison: SET-R/Healthy Home vs Treatment As Usual (TAU); To determine sample size for the grant proposal we conducted simulation studies in Mplus (Muthén & Muthén, 2010) following the procedure described by Muthén and Muthén (2002). Each simulation created 10,000 datasets, assuming a medium-size (d = .5) intervention effect, and attrition of 10% at each assessment. For α= .05, the power estimate was at or above 80% with a sample of 172 mothers; Test type: Superiority; p < .05, Generalized Estimating Equations (GEE); GEE allowed the examination of trajectories from baseline through the 12 month follow-up; Slope = -0.24, Standard Error of Mean 0.11

2. Primary Outcome: Trajectory of Anxiety of Participants
Description: Self-reported experience with anxiety symptoms as measured by the PROMIS anxiety scale over the past 7 days. Each item is scored 1-5 (1 = Never; 5 = Always), yielding a total between 8 and 40.
Time Frame: baseline, 4, 8 and 12 months
Population: Intent to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Number analyzed (Participants) | 85 | 87
Participants
  Participants Above Clinical Cutoff: Baseline | 49 | 48
  Participants Above Clinical Cutoff: 4 month | 37 | 36
  Participants Above Clinical Cutoff: 8 month | 32 | 31
  Participants Above Clinical Cutoff: 12 month | 26 | 32

3. Secondary Outcome: Trajectory of Sleep Disturbance of Participants
Description: Self-reported experience with sleep disturbance over the past 7 days as measured by the PROMIS 29 sleep disturbance subscale . Each item is scored 1-5, yielding a total between 4 and 20.
Time Frame: baseline, 4, 8 and 12 months
Population: Intent to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Number analyzed (Participants) | 85 | 87
Participants
  Participants Above Clinical Cutoff: Baseline | 30 | 28
  Participants Above Clinical Cutoff: 4 month | 24 | 17
  Participants Above Clinical Cutoff: 8 month | 16 | 25
  Participants Above Clinical Cutoff: 12 month | 13 | 19

4. Secondary Outcome: Trajectory of Fatigue of Participants
Description: Self-reported experience with fatigue over the past 7 days as measured by the PROMIS 29 fatigue subscale. Each item is scored 1-5, yielding a total between 5 and 20.
Time Frame: baseline, 4, 8 and 12 months
Population: Intent to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Number analyzed (Participants) | 85 | 87
Participants
  Participants Above Clinical Cutoff: Baseline | 25 | 27
  Participants Above Clinical Cutoff: 4 month | 20 | 24
  Participants Above Clinical Cutoff: 8 month | 24 | 18
  Participants Above Clinical Cutoff: 12 month | 16 | 20

5. Secondary Outcome: Trajectory of Pain Experienced by Participants
Description: Self-reported experience with pain over the past 7 days as measured by the PROMIS 29 pain subscale. Each item is scored 1-5, yielding a total between 5 and 25.
Time Frame: baseline, 4, 8 and 12 months
Population: Intent to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Number analyzed (Participants) | 85 | 87
Participants
  Participants Above Clinical Cutoff: Baseline | 24 | 30
  Participants Above Clinical Cutoff: 4 month | 18 | 26
  Participants Above Clinical Cutoff: 8 month | 19 | 21
  Participants Above Clinical Cutoff: 12 month | 17 | 24

6. Secondary Outcome: Trajectory of Physical Function of Participants
Description: Self-reported physical function over the past 7 days as measured by the PROMIS 29 physical function subscale. Each item is scored 1-5, yielding a total between 4 and 20, with higher scores indicating better physical function.
Time Frame: baseline, 4, 8 and 12 months
Population: Intent to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Number analyzed (Participants) | 85 | 87
Participants
  Participants Better than Clinical Cutoff: Baseline | 65 | 65
  Participants Better than Clinical Cutoff: 4 month | 51 | 48
  Participants Better than Clinical Cutoff: 8 month | 50 | 53
  Participants Better than Clinical Cutoff: 12 month | 58 | 49

7. Secondary Outcome: Trajectory of Oral Health Problems of Participants
Description: Self-reported oral health as measured by the Oral Health Impact Profile. Each item is scored 1-5, yielding a total between 14 and 70.
Time Frame: baseline, 4, 8 and 12 months
Population: Intent to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Number analyzed (Participants) | 85 | 87
Participants
  Participants with More than 2 Problems: Baseline | 44 | 45
  Participants with More than 2 Problems: 4 month | 33 | 33
  Participants with More than 2 Problems: 8 month | 30 | 28
  Participants with More than 2 Problems: 12 month | 26 | 19

8. Secondary Outcome: Trajectory of Daily Smoking of Participants
Description: Self-reported Daily Smoking as measured by the Addiction Severity Index.
Time Frame: baseline, 4, 8 and 12 months
Population: Intent to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Number analyzed (Participants) | 85 | 87
Participants
  Participants who smoked in last 30 days: Baseline | 21 | 21
  Participants who smoked in last 30 days: 4 month | 16 | 17
  Participants who smoked in last 30 days: 8 month | 16 | 16
  Participants who smoked in last 30 days: 12 month | 14 | 18

9. Secondary Outcome: Trajectory of Alcohol Intoxication of Participants
Description: Self-reported Alcohol Intoxication as measured by the Addiction Severity Index.
Time Frame: baseline, 4, 8 and 12 months
Population: Intent to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Number analyzed (Participants) | 85 | 87
Participants
  Number intoxicated in last 30 days: Baseline | 4 | 3
  Number intoxicated in last 30 days: 4 month | 4 | 4
  Number intoxicated in last 30 days: 8 month | 7 | 4
  Number intoxicated in last 30 days: 12 month | 4 | 7

10. Secondary Outcome: Trajectory of Illicit Drug Use of Participants
Description: Self-reported Illicit Drug Use as measured by the Addiction Severity Index.
Time Frame: baseline, 4, 8 and 12 months
Population: Intent to Treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
Number analyzed (Participants) | 85 | 87
Participants
  Number who used drugs in last 30 days: Baseline | 12 | 8
  Number who used drugs in last 30 days: 4 month | 7 | 5
  Number who used drugs in last 30 days: 8 month | 7 | 3
  Number who used drugs in last 30 days: 12 month | 9 | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | SET-R/Healthy Home | Treatment As Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/87
Other Adverse Events (participants affected / at risk) | 0/86 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT02702193/Prot_SAP_000.pdf